CLINICAL TRIAL: NCT02328131
Title: European Registry on the Management of Helicobacter Pylori Infection
Status: Recruiting | Type: Observational
Sponsor: Javier P. Gisbert (Other)
Responsible Party: Sponsor-Investigator, Javier P. Gisbert, Javier P. Gisbert MD, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Other Study IDs: Hp-EuReg
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The great diversity of regimens and treatment lines, the different efficacy of these, mostly due to the increase in bacterial antibiotic resistance and regional differences, requires a continuous critical analysis of clinical practice, evaluating systematically the efficacy and safety of the different regimens and the cost-effectiveness of the different diagnostic-therapeutic strategies. This will help in the design of an efficient and optimized treatment that will reduce number of re-treatments, diagnostic tests and the appearance of associated pathologies such as peptic ulcers, gastrointestinal bleeding and, probably, gastric cancers. Therefore, the evaluation of real clinical practice using non-interventionist registries will help to improve the design and organization of European Consensus on the management of H. pylori infection, which is the best way to establish healthcare efficiency.

Primary aim

To obtain a database registering systematically over a year a large and representative sample of routine clinical practice of European gastroenterologists in order to produce descriptive studies of the management of H. pylori infection.

Secondary aims

1. To evaluate H. pylori infection consensus and clinical guidelines implementation in different countries.
2. To perform studies focused on epidemiology, efficacy and safety of the commonly used treatments to eradicate H. pylori.
3. To evaluate accessibility to healthcare technologies and drugs used in the management of H. pylori infection.
4. To allow the development of partial and specific analysis by the participating researchers after approval by the Registry's Scientific Committee

Methodology Non-interventionist prospective multicentre international registry promoted by the European Helicobacter Study Group. A renowned gastroenterologist from each country was selected as Local Coordinator (30 countries). They will in turn select up to ten gastroenterologists per country that will register the routine clinical practice consultations they receive over 10 years in an electronic Case Report Form (e-CRF). Variables retrieved will include clinical, diagnostic, treatment, eradication confirmation and outcome data. The database will allow researchers to perform specific subanalysis after approval by the Scientific Committee of the study.

DETAILED DESCRIPTION:
Abstract

Introduction: H. pylori selectively infects the human stomach mucosa, being the most prevalent chronic infection in the world. Its prevalence correlates with socioeconomic factors and it is higher in older individuals. H. pylori presence causes chronic gastritis in 100% of infected patients and is the major cause of relevant diseases such as atrophic gastritis, peptic ulcer disease and gastric cancer; it is for this reason that from a public health standpoint it is considered a high impact pathogen, responsible of a significant morbidity and mortality. Nowadays there are Consensus and Clinical Guidelines regarding the infection management at a European level and in most of the states, but no data have shown the level of implementation of these recommendations. The high costs that this infection carries both socially and to the health system require the continuous and systematic assessment of the diagnostic and treatment strategies, as well as the accessibility to diagnostic methods and most efficient drugs.

Aim: To register the treatment, diagnosis and management strategies of H. pylori infected adult patients in the Digestive Services outpatient clinics throughout Europe.

Methods: Non-interventionist prospective multicentre international registry promoted by the European Helicobacter Study Group. A renowned gastroenterologist from each country was selected as Local Coordinator (30 countries). They will in turn select up to ten gastroenterologists per country that will register the routine clinical practice consultations they receive over 10 years in an electronic Case Report Form (e-CRF). Variables retrieved will include clinical, diagnostic, treatment, eradication confirmation and outcome data. The database will allow researchers to perform specific subanalysis after approval by the Scientific Committee of the study.

INTRODUCTION

H. pylori presence causes chronic gastritis in 100% of infected patients and is the major cause of relevant diseases such as atrophic gastritis, peptic ulcer disease and gastric cancer. H. pylori eradication prevents peptic ulcer recurrence and its complications, and decreases the incidence of gastric cancer. H. pylori eradication in patients with peptic ulcer or even functional or non-investigated dyspepsia is a cost-effective strategy.

The most common clinical manifestation of H. pylori infection is dyspepsia, a major health problem, whose prevalence reaches more than 10% among adult populations with its attendant burden of morbidity and health system costs in diagnosis and treatment. Approximately 20% to 30% of people in the community each year report chronic or recurrent dyspeptic symptoms, and consultations for dyspepsia account for up to 40% of referrals among gastroenterology outpatients, the "test-and-treat" strategy being the most cost-effective. Moreover, H. pylori is the major cause of peptic ulcer disease, causing over 90% of duodenal and 70% of gastric ulcers. Considerable evidence supports that the nature of the chronic inflammatory process driven by H. pylori is of critical importance in gastric carcinogenesis (adenocarcinoma and mucosa-associated lymphoid tissue -MALT- lymphoma). It is for that reason that the WHO's International Agency for Research on Cancer classified H. pylori as a group 1 (definite) carcinogen.

Scientific evidence demonstrates that diagnosis and eradication of H. pylori is the most cost-effective strategy in the management of dyspepsia, peptic ulcer and gastric cancer prevention. The treatment regimens are very diverse and have changed overtime. Monotherapies and treatments with two drugs did not achieve acceptable eradication rates. The commonly recommended regimen in most Consensus Conferences is the standard triple regimen, combining two antibiotics (clarithromycin with amoxicillin or metronidazole) and a proton pump inhibitor (PPI) for 7 to 14 days. Another recommended alternative is bismuth-containing quadruple therapy (PPI, tetracycline, metronidazole and bismuth salts). In the last years, results with new and efficient rescue regimens including levofloxacin have been published. Lately, new treatments have been proposed, including non-bismuth quadruple regimens, with two main variants: the "sequential" treatment (an induction phase with PPI and amoxicillin and a second phase with PPI, clarithromycin and metronidazole) and the "concomitant" treatment (same four drugs taken altogether).

The great diversity of regimens and treatment lines, the different efficacy of these, mostly due to the increase in bacterial antibiotic resistance and regional differences, requires a continuous critical analysis of clinical practice, evaluating systematically the efficacy and safety of the different regimens and the cost-effectiveness of the different diagnostic-therapeutic strategies. This will help in the design of an efficient and optimized treatment that will reduce number of re-treatments, diagnostic tests and the appearance of associated pathologies such as peptic ulcers, gastrointestinal bleeding and, probably, gastric cancers. Therefore, the evaluation of real clinical practice using non-interventionist registries will help to improve the design and organization of European Consensus on the management of H. pylori infection, which is the best way to establish healthcare efficiency.

AIMS

Primary aim To obtain a database registering systematically over a year a large and representative sample of routine clinical practice of European gastroenterologists in order to produce descriptive studies of the management of H. pylori infection.

Secondary aims

1. To evaluate H. pylori infection consensus and clinical guidelines implementation in different countries.
2. To perform studies focused on epidemiology, efficacy and safety of the commonly used treatments to eradicate H. pylori.
3. To evaluate accessibility to healthcare technologies and drugs used in the management of H. pylori infection.
4. To allow the development of partial and specific analysis by the participating researchers after approval by the Registry's Scientific Committee.

METHODS

International multicenter prospective non-interventionist registry promoted by the European Helicobacter Study Group.

Scientific Committee

* Javier P. Gisbert (President)
* Francis Megraud
* Colm O'Morain
* Adrian G. McNicholl

Local Coordinators

A list of European Countries has been selected. Included countries were those having at least ten clinical research publications in PubMed regarding H. pylori infection.

In each country a Local Coordinator was selected based on its clinical and research activity (Table I).

The Local Coordinators will constitute the monitoring and drafting committee of the registry.

The Local Coordinators will be in charge of selecting up to 10 recruiting investigators in each country and will be in charge of the follow up and quality of the recruiting; they will be the link between promoters and recruiting investigators.

Recruiter Investigators

The Recruiting Investigators must be gastroenterologists attending an adult population with a gastroenterology outpatient clinic that assists H. pylori infected patients. Before acceptance the outpatient clinic must attend, in a clinical routine basis, patients in which H. pylori diagnosis or treatment is indicated. Eradication confirmation tests have to be performed routinely. They will register the study variables of their own routine clinical practice in an e-CRF.

Study Variables

Anonymised Patient Identifiers

* Country/Centre/Investigator
* Autonumeric Patient identifier number
* Gender
* Date of Birth
* Ethnic Background History and Comorbidity
* Drug allergies
* Relevant comorbidities
* Current concomitant medication Data on Infection
* Indication for diagnosis and treatment
* Upper Gastrointestinal tract symptoms
* Diagnostic Test for current treatment
* Number and type of previous eradication attempts Prescribed Treatment
* Drugs
* Dosage and intakes per day
* Length of treatment Compliance
* Adherence to treatment (yes/no >90%) Adverse Events
* Type of event, intensity, duration and relation with treatment
* Treatment withdrawal due to adverse events. Efficacy
* Eradication (yes/no), test used, and date

ELIGIBILITY:
Inclusion Criteria:

* Infected adult patients by Helicobacter pylori

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infected adult patients by Helicobacter pylori
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-06; Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Prescribed treatment for H. pylori | 1 year
  * Drugs
  * Dosage and intakes
  * Length of treatment

SECONDARY OUTCOMES:
Adverse Events | 1 year
  * Type, intensity, duration and relation with treatment
  * Treatment withdrawal due to adverse event
Efficacy of treatment | 1 year
  Eradication (yes/no), test used and date
Anonymised patient identifiers | 1 year
  * Country/Centre/Investigator
  * Autonumeric Patient identifier number
  * Gender
  * Date of Birth
  * Ethnic Background

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pérez Gisbert, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (30):
- Medical University Wien, Vienna, Austria
- CHU de Charleroi, Charleroi, Charleroi, Belgium
- Medical University of Sofia, Sofia, Bulgaria
- University Hospital Merkur, Zagreb, Croatia
- Charles University Faculty of Medicine, Prague, Czechia
- Køge University Hospital, Køge, Denmark
- University of Tartu, Tartu, Estonia
- Herttoniemi Hospital, Helsinki, Helsinki, Finland
- Hôpital Pellegrin, Bordeaux, France
- Medizin Uni Magdeburg, Magdeburg, Germany
- Gastroenterology Clinic, Henry Dunant Hospital, Athens, Greece
- Ferencváros Health Centre, Gaastroenterology, Budapest, Hungary
- Adelaide Meath Hospital, Dublin, Dublin, Ireland
- Studio Gasbarrini, Roma, Italy
- Digestive Diseases Centre GASTRO, Riga, Latvia
- Lithuanian university of Health Sciences Hospital, Kaunas, Lithuania
- Ikazia Ziekenhuis/ Erasmus Medisch Centrum, Rotterdam, Netherlands
- Central Hospital of Ostfold, Fredrikstad, Norway
- Departament of Gastroenterology, Medical Centre for Postgraduate Education, Warsaw, Poland
- Porto, Porto, Portugal
- Timisoara, Timișoara, Romania
- Central Scientific Research Institute of Gastroenterology, Moscow, Russia
- Clinical Center of Serbia, Belgrade, Serbia
- DC Rogaska, Rogaška Slatina, Slovenia
- Hospital de La Princesa, Madrid, Madrid, Spain
- Uppsala University Hospital., Uppsala, Sweden
- University Hospital Basel, Basel, Switzerland
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)
- National Medical University, Kiev, Ukraine
- Leeds General Infirmiry Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arkkila PE, Seppala K, Kosunen TU, Sipponen P, Makinen J, Rautelin H, Farkkila M. Helicobacter pylori eradication as the sole treatment for gastric and duodenal ulcers. Eur J Gastroenterol Hepatol. 2005 Jan;17(1):93-101. doi: 10.1097/00042737-200501000-00018. PMID 15647648
- [Background] Azevedo NF, Huntington J, Goodman KJ. The epidemiology of Helicobacter pylori and public health implications. Helicobacter. 2009 Sep;14 Suppl 1:1-7. doi: 10.1111/j.1523-5378.2009.00703.x. PMID 19712161
- [Background] Broutet N, Tchamgoue S, Pereira E, Lamouliatte H, Salamon R, Megraud F. Risk factors for failure of Helicobacter pylori therapy--results of an individual data analysis of 2751 patients. Aliment Pharmacol Ther. 2003 Jan;17(1):99-109. doi: 10.1046/j.1365-2036.2003.01396.x. PMID 12492738
- [Background] de Vries AC, van Grieken NC, Looman CW, Casparie MK, de Vries E, Meijer GA, Kuipers EJ. Gastric cancer risk in patients with premalignant gastric lesions: a nationwide cohort study in the Netherlands. Gastroenterology. 2008 Apr;134(4):945-52. doi: 10.1053/j.gastro.2008.01.071. Epub 2008 Jan 30. PMID 18395075
- [Background] Ford A, Moayyedi P. How can the current strategies for Helicobacter pylori eradication therapy be improved? Can J Gastroenterol. 2003 Jun;17 Suppl B:36B-40B. doi: 10.1155/2003/714124. PMID 12845349
- [Background] Ford AC, Axon AT. Epidemiology of Helicobacter pylori infection and public health implications. Helicobacter. 2010 Sep;15 Suppl 1:1-6. doi: 10.1111/j.1523-5378.2010.00779.x. PMID 21054646
- [Background] Gisbert JP, Calvet X. Review article: the effectiveness of standard triple therapy for Helicobacter pylori has not changed over the last decade, but it is not good enough. Aliment Pharmacol Ther. 2011 Dec;34(11-12):1255-68. doi: 10.1111/j.1365-2036.2011.04887.x. Epub 2011 Oct 21. PMID 22017749
- [Background] Gisbert JP, Calvet X, O'Connor A, Megraud F, O'Morain CA. Sequential therapy for Helicobacter pylori eradication: a critical review. J Clin Gastroenterol. 2010 May-Jun;44(5):313-25. doi: 10.1097/MCG.0b013e3181c8a1a3. PMID 20054285
- [Background] Gisbert JP, Calvet X. Review article: non-bismuth quadruple (concomitant) therapy for eradication of Helicobater pylori. Aliment Pharmacol Ther. 2011 Sep;34(6):604-17. doi: 10.1111/j.1365-2036.2011.04770.x. Epub 2011 Jul 11. PMID 21745241
- [Background] Gisbert JP, Khorrami S, Carballo F, Calvet X, Gene E, Dominguez-Munoz JE. H. pylori eradication therapy vs. antisecretory non-eradication therapy (with or without long-term maintenance antisecretory therapy) for the prevention of recurrent bleeding from peptic ulcer. Cochrane Database Syst Rev. 2004;(2):CD004062. doi: 10.1002/14651858.CD004062.pub2. PMID 15106235
- [Background] Graham DY, Rimbara E. Understanding and appreciating sequential therapy for Helicobacter pylori eradication. J Clin Gastroenterol. 2011 Apr;45(4):309-13. doi: 10.1097/MCG.0b013e31820ac05e. PMID 21389810
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Greenberg ER, Anderson GL, Morgan DR, Torres J, Chey WD, Bravo LE, Dominguez RL, Ferreccio C, Herrero R, Lazcano-Ponce EC, Meza-Montenegro MM, Pena R, Pena EM, Salazar-Martinez E, Correa P, Martinez ME, Valdivieso M, Goodman GE, Crowley JJ, Baker LH. 14-day triple, 5-day concomitant, and 10-day sequential therapies for Helicobacter pylori infection in seven Latin American sites: a randomised trial. Lancet. 2011 Aug 6;378(9790):507-14. doi: 10.1016/S0140-6736(11)60825-8. Epub 2011 Jul 21. PMID 21777974
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Is there a benefit to extending the duration of Helicobacter pylori sequential therapy to 14 days? Helicobacter. 2011 Apr;16(2):146-52. doi: 10.1111/j.1523-5378.2011.00829.x. PMID 21435093
- [Background] Ikenberry SO, Harrison ME, Lichtenstein D, Dominitz JA, Anderson MA, Jagannath SB, Banerjee S, Cash BD, Fanelli RD, Gan SI, Shen B, Van Guilder T, Lee KK, Baron TH; ASGE STANDARDS OF PRACTICE COMMITTEE. The role of endoscopy in dyspepsia. Gastrointest Endosc. 2007 Dec;66(6):1071-5. doi: 10.1016/j.gie.2007.07.007. Epub 2007 Oct 29. No abstract available. PMID 18028927
- [Background] Maconi G, Sainaghi M, Molteni M, Bosani M, Gallus S, Ricci G, Alvisi V, Porro GB. Predictors of long-term outcome of functional dyspepsia and duodenal ulcer after successful Helicobacter pylori eradication--a 7-year follow-up study. Eur J Gastroenterol Hepatol. 2009 Apr;21(4):387-93. doi: 10.1097/MEG.0b013e3283069db0. PMID 19182682
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] McColl KE. Clinical practice. Helicobacter pylori infection. N Engl J Med. 2010 Apr 29;362(17):1597-604. doi: 10.1056/NEJMcp1001110. No abstract available. PMID 20427808
- [Background] McNicholl AG, Linares PM, Nyssen OP, Calvet X, Gisbert JP. Meta-analysis: esomeprazole or rabeprazole vs. first-generation pump inhibitors in the treatment of Helicobacter pylori infection. Aliment Pharmacol Ther. 2012 Sep;36(5):414-25. doi: 10.1111/j.1365-2036.2012.05211.x. Epub 2012 Jul 15. PMID 22803691
- [Background] Moayyedi P. The health economics of Helicobacter pylori infection. Best Pract Res Clin Gastroenterol. 2007;21(2):347-61. doi: 10.1016/j.bpg.2006.11.004. PMID 17382282
- [Background] Moayyedi P, Deeks J, Talley NJ, Delaney B, Forman D. An update of the Cochrane systematic review of Helicobacter pylori eradication therapy in nonulcer dyspepsia: resolving the discrepancy between systematic reviews. Am J Gastroenterol. 2003 Dec;98(12):2621-6. doi: 10.1111/j.1572-0241.2003.08724.x. PMID 14687807
- [Background] Niv Y, Hazazi R. Helicobacter pylori recurrence in developed and developing countries: meta-analysis of 13C-urea breath test follow-up after eradication. Helicobacter. 2008 Feb;13(1):56-61. doi: 10.1111/j.1523-5378.2008.00571.x. PMID 18205667
- [Background] Oderda G, Shcherbakov P, Bontems P, Urruzuno P, Romano C, Gottrand F, Gomez MJ, Ravelli A, Gandullia P, Roma E, Cadranel S, De Giacomo C, Canani RB, Rutigliano V, Pehlivanoglu E, Kalach N, Roggero P, Celinska-Cedro D, Drumm B, Casswall T, Ashorn M, Arvanitakis SN; European Pediatric Task Force on Helicobacter pylori. Results from the pediatric European register for treatment of Helicobacter pylori (PERTH). Helicobacter. 2007 Apr;12(2):150-6. doi: 10.1111/j.1523-5378.2007.00485.x. PMID 17309752
- [Background] Rokkas T, Sechopoulos P, Robotis I, Margantinis G, Pistiolas D. Cumulative H. pylori eradication rates in clinical practice by adopting first and second-line regimens proposed by the Maastricht III consensus and a third-line empirical regimen. Am J Gastroenterol. 2009 Jan;104(1):21-5. doi: 10.1038/ajg.2008.87. PMID 19098844
- [Derived] Nyssen OP, Ortega GJ, Jonaitis L, Perez-Aisa A, Tepes B, Lucendo AJ, Tejedor-Tejada J, Bumane R, Garre A, Huguet JM, Perona M, Nunez O, Pabon-Carrasco M, Castro-Fernandez M, Areia M, Barrio J, Loro AM, Butler TJ, Marcos MS, Keco-Huerga A, Cajal MD, Denkovski M, Pavoni M, Buzas GM, Lerang F, Losurdo G, Wolfe Garcia PM, Phull PS, Martinez-Dominguez SJ, Kupcinskas J, Leja M, Marcos-Pinto R, Smith SM, Gasbarrini A, Papp V, Rodriguez BJG, Alonso MS, Villarroya RP, Mejide PP, Jimenez-Moreno M, Pascual-Mato M, Bravo-Pache C, Montes M, Cano-Catala A, Parra P, Moreira L, Megraud F, O'Morain C, Bujanda L, Gisbert JP; Hp-EuReg investigators. Long-Term Effect of Macrolides on Helicobacter pylori Eradication: Data From the European Registry on Helicobacter pylori Management (Hp-EuReg). Helicobacter. 2026 Jan-Feb;31(1):e70107. doi: 10.1111/hel.70107. PMID 41656747
- [Derived] Tepes B, Denkovski M, Jurecic NB, Tepes K, Cano-Catala A, Parra P, Moreira L, Nyssen OP, Megraud F, O'Morain C, Gisbert JP. Second- and Third-Line Therapies for Helicobacter pylori Eradication in Slovenia: Data From 2013-2023 of the European Registry on H. pylori Management. Helicobacter. 2025 Sep-Oct;30(5):e70085. doi: 10.1111/hel.70085. PMID 41168889
- [Derived] Tepes B, Jurecic NB, Denkovski M, Vujasinovic M, Kikec Z, Bednarik J, Tepes K, Cano-Catala A, Parra P, Moreira L, Nyssen OP, Megraud F, O'Morain C, Gisbert JP. First-Line Therapy for Helicobacter pylori in Slovenia: Data From 2013 to 2023 of the European Registry on H. pylori Management. Helicobacter. 2025 Mar-Apr;30(2):e70029. doi: 10.1111/hel.70029. PMID 40178062
- [Derived] Tejedor-Tejada J, Martinez-Dominguez SJ, Hernandez L, Cano-Catala A, Parra P, Moreira L, Nyssen OP, Gisbert JP; Hp-EuReg Investigators. Management of Helicobacter pylori Infection in Spain Beyond the Data Collected in the European Registry on H. pylori Management (Hp-EuReg): Results of a Nationwide Survey. Helicobacter. 2025 Mar-Apr;30(2):e70028. doi: 10.1111/hel.70028. PMID 40167351
- [Derived] Casas Deza D, Alcedo J, Lafuente M, Lopez FJ, Perez-Aisa A, Pavoni M, Tepes B, Jonaitis L, Castro-Fernandez M, Pabon-Carrasco M, Keco-Huerga A, Voynovan I, Bujanda L, Lucendo AJ, Brglez Jurecic N, Denkovski M, Vologzanina L, Rodrigo L, Martinez-Dominguez SJ, Fadieienko G, Huguet JM, Abdulkhakov R, Abdulkhakov SR, Alcaide N, Velayos B, Hernandez L, Bordin DS, Gasbarrini A, Kupcinskas J, Babayeva G, Gridnyev O, Leja M, Rokkas T, Marcos-Pinto R, Lerang F, Boltin D, Mestrovic A, Smith SM, Venerito M, Boyanova L, Milivojevic V, Doulberis M, Kunovsky L, Parra P, Cano-Catala A, Moreira L, Nyssen OP, Megraud F, Morain CO, Gisbert JP; Hp-EuReg investigators. Probiotics Prescribed With Helicobacter pylori Eradication Therapy in Europe: Usage Pattern, Effectiveness, and Safety. Results From the European Registry on Helicobacter pylori Management (Hp-EuReg). Am J Gastroenterol. 2025 Nov 1;120(11):2644-2659. doi: 10.14309/ajg.0000000000003351. Epub 2025 Feb 4. PMID 39902822
- [Derived] Olmedo L, Calvet X, Gene E, Bordin DS, Voynovan I, Castro-Fernandez M, Pabon-Carrasco M, Keco-Huerga A, Perez-Aisa A, Lucendo AJ, Rodrigo L, Sarsenbaeva AS, Khlinov IB, Fadieienko G, Zaytsev O, Lanas A, Martinez-Dominguez SJ, Alfaro E, Jonaitis L, Nunez O, Pellicano R, Hernandez L, Gridnyev O, Kupcinskas J, Gasbarrini A, Boltin D, Niv Y, Babayeva G, Marcos-Pinto R, Tepes B, Venerito M, Papp V, Lerang F, Leja M, Phull PS, Marlicz W, Doulberis M, Smith SM, Milivojevic V, Kunovsky L, Mestrovic A, Matysiak-Budnik T, Simsek H, Cano-Catala A, Puig I, Moreira L, Parra P, Nyssen OP, Megraud F, O'Morain C, Gisbert JP; Hp-EuReg investigators*. Evolution of the use, effectiveness and safety of bismuth-containing quadruple therapy for Helicobacter pylori infection between 2013 and 2021: results from the European registry on H. pylori management (Hp-EuReg). Gut. 2024 Dec 10;74(1):15-25. doi: 10.1136/gutjnl-2024-332804. PMID 39461739
- [Derived] Martinez-Dominguez SJ, Nyssen OP, Lanas A, Alfaro E, Jonaitis L, Mahmudov U, Voynovan I, Gulustan B, Rodrigo L, Fiorini G, Perez-Aisa A, Tejedor-Tejada J, Tepes B, Vologzanina L, Mammadov E, Lerang F, Oglu QFV, Bakulina NV, Abdulkhakov R, Tatiana I, Butler TJ, Sarsenbaeva AS, Bumane R, Lucendo AJ, Romano M, Bujanda L, Abdulkhakov SR, Zaytsev O, Pabon-Carrasco M, Keco-Huerga A, Denkovski M, Huguet JM, Perona M, Nunez O, Pavoni M, Fadieienko G, Alekseenko S, Smith SM, Hernandez L, Kupcinskas J, Bordin DS, Leja M, Gasbarrini A, Gridnyev O, Cano-Catala A, Parra P, Moreira L, Megraud F, O'Morain C, Gisbert JP; Hp-EuReg Investigators. Indications of Helicobacter pylori Eradication Treatment and Its Influence on Prescriptions and Effectiveness (Hp-EuReg). Helicobacter. 2024 Jul-Aug;29(4):e13111. doi: 10.1111/hel.13111. PMID 39001621
- [Derived] Bujanda L, Nyssen OP, Ramos J, Bordin DS, Tepes B, Perez-Aisa A, Pavoni M, Castro-Fernandez M, Lerang F, Leja M, Rodrigo L, Rokkas T, Kupcinskas J, Jonaitis L, Shvets O, Gasbarrini A, Simsek H, Phull PS, Buzas GM, Machado JC, Boltin D, Boyanova L, Tonkic A, Marlicz W, Venerito M, Vologzanina L, Fadieienko GD, Fiorini G, Resina E, Munoz R, Cano-Catala A, Puig I, Garcia-Morales N, Hernandez L, Moreira L, Megraud F, Morain CO, Montes M, Gisbert JP; Hp-EuReg investigators; Hp-EuReg investigators. Effectiveness of Helicobacter pylori Treatments According to Antibiotic Resistance. Am J Gastroenterol. 2024 Apr 1;119(4):646-654. doi: 10.14309/ajg.0000000000002600. Epub 2023 Nov 17. PMID 37983769
- [Derived] Burgos-Santamaria D, Nyssen OP, Gasbarrini A, Vaira D, Perez-Aisa A, Rodrigo L, Pellicano R, Keco-Huerga A, Pabon-Carrasco M, Castro-Fernandez M, Boltin D, Barrio J, Phull P, Kupcinskas J, Jonaitis L, Ortiz-Polo I, Tepes B, Lucendo AJ, Huguet JM, Areia M, Jurecic NB, Denkovski M, Bujanda L, Ramos-San Roman J, Cuadrado-Lavin A, Gomez-Camarero J, Jimenez Moreno MA, Lanas A, Martinez-Dominguez SJ, Alfaro E, Marcos-Pinto R, Milivojevic V, Rokkas T, Leja M, Smith S, Tonkic A, Buzas GM, Doulberis M, Venerito M, Lerang F, Bordin DS, Lamy V, Capelle LG, Marlicz W, Dobru D, Gridnyev O, Puig I, Megraud F, O'Morain C, Gisbert JP; Hp-EuReg Investigators. Empirical rescue treatment of Helicobacter pylori infection in third and subsequent lines: 8-year experience in 2144 patients from the European Registry on H. pylori management (Hp-EuReg). Gut. 2022 Dec 5:gutjnl-2022-328232. doi: 10.1136/gutjnl-2022-328232. Online ahead of print. PMID 36591610
- [Derived] Nyssen OP, Vaira D, Perez Aisa A, Rodrigo L, Castro-Fernandez M, Jonaitis L, Tepes B, Vologzhanina L, Caldas M, Lanas A, Lucendo AJ, Bujanda L, Ortuno J, Barrio J, Huguet JM, Voynovan I, Lasala JP, Sarsenbaeva AS, Fernandez-Salazar L, Molina-Infante J, Jurecic NB, Areia M, Gasbarrini A, Kupcinskas J, Bordin D, Marcos-Pinto R, Lerang F, Leja M, Buzas GM, Niv Y, Rokkas T, Phull P, Smith S, Shvets O, Venerito M, Milivojevic V, Simsek I, Lamy V, Bytzer P, Boyanova L, Kunovsky L, Beglinger C, Doulberis M, Marlicz W, Goldis A, Tonkic A, Capelle L, Puig I, Megraud F, Morain CO, Gisbert JP; European Registry on Helicobacter pylori Management Hp-EuReg Investigators. Empirical Second-Line Therapy in 5000 Patients of the European Registry on Helicobacter pylori Management (Hp-EuReg). Clin Gastroenterol Hepatol. 2022 Oct;20(10):2243-2257. doi: 10.1016/j.cgh.2021.12.025. Epub 2021 Dec 23. PMID 34954341
- [Derived] Nyssen OP, Perez-Aisa A, Tepes B, Castro-Fernandez M, Kupcinskas J, Jonaitis L, Bujanda L, Lucendo A, Jurecic NB, Perez-Lasala J, Shvets O, Fadeenko G, Huguet JM, Kikec Z, Bordin D, Voynovan I, Leja M, Machado JC, Areia M, Fernandez-Salazar L, Rodrigo L, Alekseenko S, Barrio J, Ortuno J, Perona M, Vologzhanina L, Romero PM, Zaytsev O, Rokkas T, Georgopoulos S, Pellicano R, Buzas GM, Modolell I, Gomez Rodriguez BJ, Simsek I, Simsek C, Lafuente MR, Ilchishina T, Camarero JG, Dominguez-Cajal M, Ntouli V, Dekhnich NN, Phull P, Nunez O, Lerang F, Venerito M, Heluwaert F, Tonkic A, Caldas M, Puig I, Megraud F, O'Morain C, Gisbert JP; Hp-EuReg Investigators. Adverse Event Profile During the Treatment of Helicobacter pylori: A Real-World Experience of 22,000 Patients From the European Registry on H. pylori Management (Hp-EuReg). Am J Gastroenterol. 2021 Jun 1;116(6):1220-1229. doi: 10.14309/ajg.0000000000001246. PMID 33840725
- [Derived] Nyssen OP, Perez-Aisa A, Castro-Fernandez M, Pellicano R, Huguet JM, Rodrigo L, Ortun J, O, Gomez-Rodriguez BJ, Pinto RM, Areia M, Perona M, Nunez O, Romano M, Gravina AG, Pozzati L, Fernandez-Bermejo M, Venerito M, Malfertheiner P, Fernanadez-Salazar L, Gasbarrini A, Vaira D, Puig I, Megraud F, O'Morain C, Gisbert JP; Hp-EuReg investigators. European Registry on Helicobacter pylori management: Single-capsule bismuth quadruple therapy is effective in real-world clinical practice. United European Gastroenterol J. 2021 Feb;9(1):38-46. doi: 10.1177/2050640620972615. Epub 2021 Feb 11. PMID 33176617
- [Derived] McNicholl AG, Bordin DS, Lucendo A, Fadeenko G, Fernandez MC, Voynovan I, Zakharova NV, Sarsenbaeva AS, Bujanda L, Perez-Aisa A, Vologzhanina L, Zaytsev O, Ilchishina T, Coba C, Lasala JP, Alekseenko S, Modolell I, Molina-Infante J, Ruiz-Zorrilla Lopez R, Alonso-Galan H, Moreno NF, Hinojosa J, Santaella I, Varela P, Gonzalez-Cordero PL, Barrio J, Dominguez-Jimenez JL, Nunez O, Alcedo J, Nyssen OP, Caldas M, Donday MG, Shvetz O, Megraud F, O'Morain C, Gisbert JP. Combination of Bismuth and Standard Triple Therapy Eradicates Helicobacter pylori Infection in More than 90% of Patients. Clin Gastroenterol Hepatol. 2020 Jan;18(1):89-98. doi: 10.1016/j.cgh.2019.03.048. Epub 2019 Apr 10. PMID 30978536